CLINICAL TRIAL: NCT00001938
Title: A Pilot Study of Proteomic Evaluation of Epithelial Ovarian Cancer Patients in First Clinical Remission: Development of a Protein Fingerprint Profile Associated With Relapse
Brief Title: A Pilot Study of a Protein Profile Test in Ovarian Cancer Patients in Remission to See if Protein Changes Can Predict Relapse (be Predictive of Cancer Relapse)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000018; 00-C-0018; NCT00020033 (obsolete NCT alias)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Neoplasm
Keywords: Ovarian Cancer; Proteomics
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine, pleural/peritoneal fluid, tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Every cell in the human body contains hundreds of thousands of genes and the proteins made by the genes. Sometimes changes take place in the genes or proteins that may make the cells more likely to develop into cancer. An experimental protein profile test that finds these changes may be able to provide information about whose cancer will stay in remission and whose will return.

Volunteer patients whose epithelial ovarian cancer is in remission are eligible for this study. Specimens will be collected from blood, saliva, and urine for the first protein profile test. Sample sets for more protein profile tests will be collected at follow-up visits 1 month and 3 months later and every 3 months afterward. If and when the cancer returns, an additional sample set will be obtained and a biopsy of the relapsed tumor will be taken both for a protein profile test and for review of the function and structure of the disease (pathology review). The protein profiles from these samples will be compared to those samples already collected to detect protein pattern changes. The amount of lysophosphatidic acid (LPA) in the blood, a sign of ovarian cancer, will also be measured to see if LPA is useful in detecting the return of ovarian cancer.

If patients get fluid in the stomach or chest, it will be tested for cancer cells and proteins made by the tumor. If a physical exam or CT scan indicates a possible return of the cancer, a biopsy will be performed and a sample saved for a protein profile.

DETAILED DESCRIPTION:
Over 80 percent of advanced stage epithelial cancer patients relapse after attaining first clinical remission with standard platinum/paclitaxel-based chemotherapy. Surrogate biomarkers are needed for the evaluation of efficacy of treatment and for use as predictors of disease in screening and for relapse diagnosis. CA-125, the existing ovarian cancer marker, will become elevated with relapse in some but not all of the 80 percent of patients for whom it was increased at initial diagnosis. Elevation in CA-125 may precede clinical evidence of relapse by as much as 6 - 10 months or lag behind clinical relapse by the same time intervals, making it a less than satisfactory clinical tool. Emerging proteomic technologies allow for scanning of cellular proteins in a simple, short, reproducible, and quantitative chemical assay. We hypothesize that changes in a patient s protein pattern will be detectable and will be reliably associated with relapse. This protocol is a pilot study for our ability to ascertain and evaluate samples from ovarian cancer patients followed in first clinical remission, and investigate whether analysis of sequential protein fingerprints will yield a reproducible pattern of change that may be associated with relapse.

ELIGIBILITY:
* INCLUSION CRITERIA

All patients in first clinical remission from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma or stage IIC clear cell histology epithelial ovarian cancer as defined by: normal CA-125, normal physical exam, normal post hysterectomy pelvic examination, no evidence of disease on CT scan or other noninvasive reassessment.

Entry within 9 weeks of completion of final cycle of chemotherapy (within 12 weeks of last administration of chemotherapy).

S/P completion of primary therapy with standard platinum/paclitaxel or carboplatin/paclitaxel-containing chemotherapy and in confirmed clinical complete response.

At least one block from the primary tumor must be received. (If available, a sample of frozen primary tumor should also be forwarded).

ECOG performance status of 0, 1, or 2.

EXCLUSION CRITERIA

Patients with nonepithelial ovarian cancer, or mixed epithelial/nonepithelial ovarian cancer.

Patients may not be receiving chemotherapy, hormonal therapy, alternative therapy, or radiation therapy. No therapy of any kind is allowed while the patient is on-study. Replacement hormonal therapy is not allowed.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical population of patients in first clinical remisssion from treatment of FIGO stage III/IV primary peritoneal, fallopian tube, or epithelial ovarian carcinoma or stage II clear cell histology epithelial ovarian cancer. Entry within 12 weeks of last administration of chemotherapy. S/P completion of primary therapy with standard platinum/paclitaxel or carboplatin/paclitaxel-containing chemotherapy and in inconfirmed clinical complete response.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2000-04-24 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Biomarker analysis | At 1 mo; every 3 mos; at progression or 24 mos of complete clinical remission; every 6 mos after 3 yrs on study; and annually after 5 yrs on study
  creation of protein profiles of epithelial ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Patsner B, Orr JW Jr, Mann WJ Jr, Taylor PT, Partridge E, Allmen T. Does serum CA-125 level prior to second-look laparotomy for invasive ovarian adenocarcinoma predict size of residual disease? Gynecol Oncol. 1990 Sep;38(3):373-6. doi: 10.1016/0090-8258(90)90076-w. PMID 2227551
- [Background] Woolas RP, Xu FJ, Jacobs IJ, Yu YH, Daly L, Berchuck A, Soper JT, Clarke-Pearson DL, Oram DH, Bast RC Jr. Elevation of multiple serum markers in patients with stage I ovarian cancer. J Natl Cancer Inst. 1993 Nov 3;85(21):1748-51. doi: 10.1093/jnci/85.21.1748. PMID 8411259
- [Background] Rosenthal A, Jacobs I. Ovarian cancer screening. Semin Oncol. 1998 Jun;25(3):315-25. PMID 9633843
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-C-0018.html